CLINICAL TRIAL: NCT00377130
Title: Stress Management Therapy for Patients Undergoing Chemotherapy
Brief Title: Stress Management Therapy in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCUSF 0501; SCUSF-0501 (Other: SunCoast CCOP Research Base); HLMCC-0501 (Other: H. Lee Moffitt Cancer Center Research Base); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2010-09

CONDITIONS: Cancer; Psychological Stress; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasms; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I- Usual psychological care (No Intervention): Usual psychological care- no intervention
- Self administered Stress Management (Experimental): Self-Administered Stress Management Training Plus Usual Psychosocial Care
  Interventions: Other: Self Administered Stress Management

INTERVENTIONS:
Other: Self Administered Stress Management — The SSMT kit includes a DVD and booklet will discuss the sources and manifestations of stress during chemotherapy and the potential benefits of stress management training. The videotape/DVD and booklet will also include brief instruction in paced breathing, progressive muscle relaxation with guided imagery, and use of coping self-statements as well as recommendations for practicing the techniques before the start of chemotherapy and using them after the start of treatment. The exercise combines abbreviated progressive muscle relaxation training with use of relaxing mental imagery. The "positive thinking" exercise provides participants with brief instruction in the use of coping self-statements using techniques borrowed from stress inoculation training.
  Other Names: self-administered stress management training (SSMT)
  Arms: Self administered Stress Management

SUMMARY:
RATIONALE: A stress-management program may improve quality of life and reduce anxiety and depression in patients receiving chemotherapy for cancer.

PURPOSE: This randomized clinical trial is studying how well stress management therapy works in patients receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if a self-administered stress management intervention is effective in improving quality of life and decreasing psychological distress (anxiety and depression) in Hispanic and non-Hispanic patients receiving cancer chemotherapy.

Secondary

* Determine if the degree of acculturation in Hispanics influences the observed helpfulness of the intervention.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, use of psychotropic drugs (yes vs no), and ethnicity (Hispanic vs non-Hispanic). Patients are randomized to 1 of 2 arms.

* Arm I (self-administered stress management training plus usual psychosocial care): Patients receive a video DVD, audio CD, and brochure that provides information and instruction in 3 stress management training techniques (progressive muscle relaxation training and guided imagery, abdominal breathing, and coping skills training) to use during chemotherapy. Patients also receive usual psychosocial care.
* Arm II (usual psychosocial care only): Patients receive usual psychosocial care.

Patients complete questionnaires to assess mood, quality of life, and other factors at baseline and before chemotherapy courses 2, 3, and 4.

PROJECTED ACCRUAL: A total of 442 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* At least 18 years of age
* Newly diagnosed with cancer
* Scheduled to receive a minimum of 4 cycles of intravenous chemotherapy
* Able and willing to give informed consent to participate

EXCLUSION CRITERIA:

* Had intravenous chemotherapy prior to study entry
* Are scheduled to receive radiotherapy prior to the end of the fourth cycle
* Have severe depression or other severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Quality of life | After 4th chemotherapy cycle
  Assessed at baseline (before first chemotherapy cycle) and just before the start of the second, third and fourth chemotherapy cycles.
Anxiety | after 4th chemotherapy cycle
  Assessed at baseline (before first chemotherapy cycle) and just before the start of the second, third and fourth chemotherapy cycles.
Depression | After 4th chemotherapy cycle
  Assessed at baseline (before first chemotherapy cycle) and just before the start of the second, third and fourth chemotherapy cycles.

SECONDARY OUTCOMES:
Degree of acculturation | After 4th chemotherapy cycle
  Assessed at baseline (before first chemotherapy cycle) and just before the start of the second, third and fourth chemotherapy cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Teletia Taylor, PhD, Study Chair — Howard University Cancer Center; Susan McMillan, PhD RN FAAN, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (51):
- United States (46):
  - Contra Costa Regional Medical Center, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - MBCCOP - JHS Hospital of Cook County, Chicago, Illinois
  - Savoy Medical Center, Mamou, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - William Beaumont Hospital - Troy Campus, Troy, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. John's Regional Health Center, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Dickstein Cancer Treatment Center at White Plains Hospital Center, White Plains, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center - Wilson, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Hospital East, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Mount Carmel St. Ann's Cancer Center, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - CCOP - Scott and White Hospital, Temple, Texas
  - Scott and White Cancer Institute, Temple, Texas
  - Rainier Physicians - NWMS, Puyallup, Washington
  - CCOP - Northwest, Tacoma, Washington
- Puerto Rico (5):
  - Andres Grillasca Hospital, Ponce
  - Hato Rey Hematology/Oncology Group, PSC, San Juan
  - I. Gonzalez Martinez Oncologic Hospital, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
  - San Juan City Hospital, San Juan